CLINICAL TRIAL: NCT06045104
Title: Effectiveness of Context-adapted Alternative Feeding Regimen on Recovery of Children Aged 6-59 Months From Moderate Acute Malnutrition and Uncomplicated Severe Acute Malnutrition in Bangladesh. A Cluster Randomized Control Trial
Brief Title: Alternative Feeding Regimen on Recovery of Children Aged 6-59 Months With Moderate Acute Malnutrition in Bangladesh.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Action Contre la Faim (Other); University Ghent (Other); United Nations World Food Programme (WFP) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-22128-A
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Moderate Acute Malnutrition
Keywords: Moderate Acute Malnutrition; Children; Wheat Soy Blend ++; 15 MNP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheat Soy Blend Plus Plus (WSB++) with nutrition counselling (Active Comparator): Wheat Soy Blend Plus Plus (WSB++) with nutrition counselling
  Interventions: Dietary Supplement: Wheat Soy Blend Plus Plus (WSB++) with nutrition counselling
- 15 Micro Nutrient Powder (15 MNP) with improved nutrition counselling (Experimental): 15 Micro Nutrient Powder (15 MNP) with improved nutrition counselling
  Interventions: Dietary Supplement: 15 Micro Nutrient Powder (15 MNP) with improved nutrition counselling

INTERVENTIONS:
Dietary Supplement: Wheat Soy Blend Plus Plus (WSB++) with nutrition counselling — Wheat Soy Blend Plus Plus (WSB++) with nutrition counselling
  Arms: Wheat Soy Blend Plus Plus (WSB++) with nutrition counselling
Dietary Supplement: 15 Micro Nutrient Powder (15 MNP) with improved nutrition counselling — 15 Micro Nutrient Powder (15 MNP) with improved nutrition counselling
  Arms: 15 Micro Nutrient Powder (15 MNP) with improved nutrition counselling

SUMMARY:
In spite of the large burden of acute malnutrition in the country, the Community-based Management of Acute Malnutrition (CMAM) protocol approved in Bangladesh highly deviates from the WHO normative guidance, in that it does not support the use of any currently existing nutritional products for Moderate Acute Malnutrition (MAM) cases: it relies solely on nutrition counselling. On another hand, some non-governmental organizations (NGOs) are implementing programs making a standard use of specialized nutritional products, such as nutritional supplements like Wheat Soy Blend (WSB)++ to manage MAM cases, in children of Forcibly Displaced Myanmar Nationals (FDMNs) in the refugee camps situated at the south-eastern region of the country and in some crisis-affected districts as well.

The "no-food" CMAM policy for MAM is decreasing the cost of treatment, yet this may undermine effectiveness and impact. In this context, policy makers need evidence regarding context specific, effective and scalable interventions for CMAM.

This cluster randomized control trial (cRCT) will be conducted in the host communities in Teknaf and Ukhiya sub-districts of Cox's Bazar district of Bangladesh among children aged 6-59 months suffering from MAM who will be assigned to receive either of the 2 different treatment packages for a period of 4 months (120 days). Then followed up for 6 months (180 days) post treatment completion. Each arm will consist of 280 children with MAM. Both the arms will receive nutrition counselling along with the study intervention, as follows:

In the first arm, the treatment packages for children with MAM will include a standard use of specialized nutritional products developed to address the nutritional needs of these children in acute crisis/emergency settings and widely used internationally: children with MAM will receive WSB++ with nutrition counselling for a period of 4 months (120 days),.

In the second arm, children with MAM will receive 15 MNP with improved nutrition counselling for a period of 4 months (120 days).

A cluster sampling technique will be used to enroll participants. Each Community Clinic and Union Health & Family Welfare Centers will serve as unit of cluster for the randomization.

Primary outcome variables are: 1) Daily weight gain (g/kg/d) between enrolment and end of the treatment period. 2) Recovery rate (%) at the end of the treatment period.

DETAILED DESCRIPTION:
Background

Burden:

Acute Malnutrition (AM) which is also known as 'wasting' in children under five years of age is a major and significant global health problem. It has two forms: i) Severe Acute Malnutrition [(SAM, defined as weight-for-height/length z-score (WHZ/WLZ) less than -3 standard deviations (SDs) from the median of reference population and or Mid-Upper Arm Circumference (MUAC) < 115mm, and or presence of bipedal edema)], and ii) Moderate Acute Malnutrition [(MAM, defined as WHZ/WLZ between -3SDs and <-2SDs and or MUAC ≥ 115mm to <125mm)]. It is estimated that more than half of all under five deaths are associated with undernutrition. Both MAM and SAM pose serious consequences, leading to increased morbidity and mortality, impaired intellectual development, increased risk of non-communicable diseases (NCDs) in adulthood, and suboptimal adult work capacity. Children with SAM have approximately nine times and children with MAM have approximately three times higher risk of mortality due to common communicable diseases than if they were well-nourished. A MAM child is additionally at higher risk of developing SAM if their health and nutritional condition is not monitored. The recent Lancet analysis estimated that in 2020, the COVID19 pandemic exacerbated the problem of AM with an additional 6.7 million children - equivalent to a 14.3% increase in the number of children with wasting. More than half (3.9 million) of these children would be from South Asia alone. Although prevalence of AM in many countries have reduced, still these are far from Sustainable Development Goals (SDGs) target.

Despite Bangladesh already progressed in reduction of AM by more than half between 2007 and 2017, still it has one of the highest prevalence of AM in the world. According to Bangladesh Demographic and Health Survey (BDHS) 2017 prevalence of AM under-5 children was 8.4%, while the multiple indicator cluster survey (MICS) which included a larger sample, found a slight increase from 9.6% in 2013 to 9.8% (1.5 million) in 2019. Of the total AM, 7.5% (1.1-1.2 million) were MAM. It depicts that currently in terms of reducing the prevalence of wasting among children under five to <5 %, Bangladesh has to go far away to achieve the SDG target 2.2 by 2025. It was observed that despite having recovery rate above the minimum standards of >75%, post-discharge relapse rates of AM were very high (78% for MAM 69% while 9% for SAM) in Bangladesh and Southern Ethiopia 72.1% (37.5% for MAM and 34.6% for SAM). Chang et al. 2013 found 27% (17% for MAM and 10% for SAM) relapse cases in Malawi. Therefore, after recovery and discharge a child should be followed up to assess the maintenance of the nutritional status, because it is likely that children who recovered from AM may recur as AM after returning to the same environment.

Knowledge gap:

Based on the current consensus, children with MAM should also be managed at home/community. Essential nutrition activities such as breastfeeding promotion and support, education and nutrition counselling for caregivers should be an integral part of management of children aged 6-59 months with MAM or uncomplicated SAM. WHO 19 Technical Group and Community Management of Acute Malnutrition (CMAM) Forum, 2014 recommended nutritional supplements and nutrition counselling for children with MAM. However, the latest WHO recommendation on MAM management is that it should not provide nutritional supplements routinely unless the context is highly food insecure (WHO 2017).

In Bangladesh, children with MAM receive basic medical treatment, and mothers/caregivers are provided with counselling on the use of high energy/nutrient dense local foods fortified with micronutrients in the outpatient care. Community outreach activities are given priority in promotion and support of appropriate infant and young child feeding (IYCF) practices, identification, care, referral, and follow up of children with AM.

Relevance:

In spite of the large burden of acute malnutrition in the country, the CMAM protocol approved in Bangladesh highly deviates from the WHO normative guidance, in that it does not support the use of any currently existing nutritional products for MAM cases: it relies solely on nutrition counselling. On another hand, some non-governmental organizations (NGOs) are implementing programs making a standard use of specialized nutritional supplements like Wheat Soy Blend (WSB)++ to manage MAM cases, in children of Forcibly Displaced Myanmar Nationals (FDMNs) in the refugee camps situated at the south-eastern region of the country and in some crisis-affected districts as well.

The "no-food" CMAM policy for MAM is decreasing the cost of treatment, yet this may undermine effectiveness and impact. In this context, policy makers need evidence regarding context specific, effective and scalable interventions for CMAM.

Hypothesis:

The study hypothesizes that improved nutrition counselling provided together with 15 MNP is equally effective (recovery rate) as super cereal (WSB++) in treating children aged 6-59 months with MAM for a period of 4 months (120 days).

Objectives:

Primary Objectives

1. To assess the daily weight gain and recovery rate among MAM children aged 6-59 months provided with 15 MNP with improved nutrition counselling and WSB++ with nutrition counselling provided for a period of 4 months (120 days).
2. To identify the predictors for the 'not recovered/non-responder' to the treatment(s) and regression to SAM among MAM children at the end of 4 months (120 days).

Secondary objectives

1. To evaluate the effects of nutrition counselling combined with 15 MNP and WSB++ on relapse of MAM children during a period of 6 months (180 days) post treatment (long term).
2. To evaluate the effects of nutrition counselling combined with 15 MNP and WSB++ provided solely on body composition (lean and fat mass) of MAM children at the end of 4 months (120 days) and 6 months (180 days) post treatment (long term).
3. To evaluate the effects of nutrition counselling combined with 15 MNP and WSB++ on cognitive development of MAM children at the end of 4 months (120 days) and 6 months (180 days) post treatment (long term).
4. To identify concurrent illness, and gut microbiota (in a sub-sample) at baseline and end of intervention period.
5. To evaluate the cost-effectiveness of community management of MAM children aged 6-59 months provided with nutrition counselling combined with 15 MNP and WSB++.
6. To define challenges and opportunities in scaling up the tested intervention(s) if proven to be effective alone or cost effective as well.

Methods:

Study site:

The study will be conducted in the host communities in Teknaf and Ukhiya sub-districts of Cox's Bazar district of Bangladesh.

Study Population:

This trial will be conducted in children aged 6-59 months with MAM residing in Teknaf and Ukhiya sub-districts of Cox's Bazar district of Bangladesh.

Inclusion criteria

The inclusion criteria for enrolment in the study will include:

i) Children of either sex, aged between 6-59 months having MUAC <125 mm and/or WHZ/WLZ <-2 SD ii) Absence of edema or morbidities that necessitate hospitalization iii) Children with appetite iv) Mothers/caregivers sign the consent form v) Willing to bring the child to the study site every two weeks for MAM and have a plan to stay in the community for at least next 9-10 months.

vi) Accept the intervention package and home visits for data collection and morbidity follow up.

Exclusion criteria:

The study will not include children with- i) Bipedal edema ii) MAM with clinically severe anemia, suspected tuberculosis, other chronic diseases or any congenital disorder or deformity, an ongoing episode of diarrhea, a history of persistent diarrhea in the past month.

iii) Complicated SAM cases

Study plan In this cluster randomized-controlled trial (cRCT), 560 eligible MAM children will be enrolled, treated for 4 months (120 days) and then followed up for 6 months (180 days) post treatment completion.

Study design

This cluster randomized control trial (cRCT) will include children aged 6-59 months suffering from MAM who will be assigned to receive either of the 2 different treatment packages for a period of 4 months (120 days). Then followed up for 6 months (180 days) post treatment completion. Each arm will consist of 280 children with MAM. Both the arms will receive nutrition counselling along with the study intervention, as follows:

In the first arm, the treatment packages for children with MAM will include a standard use of specialized nutritional products developed to address the nutritional needs of these children in acute crisis/emergency settings and widely used internationally: children with MAM will receive WSB++ with nutrition counselling for a period of 4 months (120 days).

In the second arm, children with MAM will receive 15 MNP with improved nutrition counselling for a period of 4 months (120 days).

Sampling technique A cluster sampling technique will be used to enroll participants. Each Community Clinic and Union Health & Family Welfare Centers will serve as unit of cluster for the randomization.

Field implementation of the interventions:

The intervention will take place in 28 community clinics (CCs) and 6 Union Health & Family Welfare Centers (UH&FWCs) in the host communities in Teknaf and Ukhiya sub-districts of Cox's Bazar district of Bangladesh. As per the national CMAM guidelines, all the participating CC/UH&FWC provides the standard care and nutrition counselling for children with MAM or uncomplicated SAM. Children with MAM from catchment areas of the selected 10 CCs/ UH&FWCs will take part in each arm. Research team, Community Health Care Providers (CHCPs), Health Assistants (HAs), Family Welfare Assistants (FWAs) and local NGO's field workers will work to conduct this study. All participating children would be receiving standard health and nutrition counselling at each occasion they attend the CCs/UH&FWC

Outcome measures/variables:

Primary effectiveness outcomes

1. Daily weight gain (g/kg/d) between enrolment and end of the treatment period (for 4 months or 120 days). If recovery was reached before the full duration of the treatment, daily weight gain will be calculated between enrolment and recovery, without stopping the treatment.
2. Recovery rate (%) at the end of the treatment period (4 months or 120 days)
3. Proportion of children free from acute malnutrition at the end of the treatment period (4 months or 120 days)

Secondary effectiveness outcomes

1. Proportion of non-response, death, defaulter and regression of MAM to SAM (among MAM children) at the end of treatment period (4 months or 120 days).
2. Incidence of relapse during a period of 6 months (180 days) post-treatment
3. Change in lean and fat mass between enrollment and end of the treatment period (4 months or 120 days) and 6 months post-treatment
4. Prevalence of concurrent infections at the end of the treatment period (4 months or 120 days) and 6 months post-treatment
5. Motor, language, and personal-social development at the end of the treatment period (4 months or 120 days) and 6 months post-treatment
6. Cost-effectiveness analysis
7. Challenges and opportunities in scaling up the tested intervention(s)
8. Feasibility and acceptability of the interventions
9. Knowledge, attitudes and practices regarding nutritional and social care of MAM

Safety outcomes

- Incidence of diarrhea, pneumonia, malaria etc. among children during study period (9-10 months)

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex, aged between 6-59 months having MUAC <125 mm and/or WHZ/WLZ <-2 SD
* Absence of edema or morbidities that necessitate hospitalization
* Children with appetite
* Mothers/caregivers sign the consent form
* Willing to bring the child to the study site every two weeks for MAM and have a plan to stay in the community for at least next 9-10 months.
* Accept the intervention package and home visits for data collection and morbidity follow up

Exclusion Criteria:

* Bipedal edema
* MAM with clinically severe anemia, suspected tuberculosis, other chronic diseases or any congenital disorder or deformity, an ongoing episode of diarrhea, a history of persistent diarrhea in the past month.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 560 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of weight gain (g/kg/d) | 4 months or 120 days
  Daily weight gain (g/kg/d) between enrolment and end of the treatment period. If recovery was reached before the full duration of the treatment, daily weight gain will be calculated between enrolment and recovery, without stopping the treatment.
Recovery rate (%) | 4 months or 120 days
  Recovery rate (%) at the end of the treatment period
Free from acute malnutrition | 4 months or 120 days
  Proportion of children free from acute malnutrition at the end of the treatment period

SECONDARY OUTCOMES:
Proportion of non-response, death, defaulter and regression of MAM to SAM | 4 months or 120 days
  Proportion of non-response, death, defaulter and regression of MAM to SAM (among MAM children) at the end of treatment period
Incidence of relapse during a period of 6 months (180 days) post-treatment | 6 months or 180 days post treatment
  Incidence of relapse during a period of 6 months (180 days) post-treatment
Change in lean and fat mass between enrollment and end of the treatment period | 4 months or 120 days) and 6 months post-treatment
  Change in lean and fat mass between enrollment and end of the treatment period
Prevalence of concurrent infections at the end of the treatment period | 4 months or 120 days) and 6 months post-treatment
  Prevalence of concurrent infections at the end of the treatment period
Motor, language, and personal-social development at the end of the treatment period | 4 months or 120 days) and 6 months post-treatment
  Motor, language, and personal-social development at the end of the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Md Munirul Islam, PhD, Principal Investigator — Scientist
Locations (1):
- Community Clinics, Teknāf, Bangladesh

IPD SHARING:
Plan to Share IPD: No